CLINICAL TRIAL: NCT02850237
Title: Pre-Hospital Cerebral Oxygenation and End-Tidal CO2 During Cardiopulmonary Resuscitation (CPR)
Acronym: CopernicusIb
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Cornelia Genbrugge, Dr., Hasselt University
Other Study IDs: CopernicusIb
Record Dates: First submitted 2016-04-20; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: out-of Hospital Cardiac Arrest
Keywords: cerebral saturation; capnography; pre-hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebral saturation will be measured pre-hospital during an out-of hospital cardiac arrest with O3TM regional oximetry for Root® (Masimo®). The O3TM regional oximetry for Root® (Masimo®) is a device that can measure not only cerebral saturation but also end-tidal CO2 (capnography). Currently, end-tidal CO2 is already measured during Advanced Life Support following most recent European Resuscitation Guidelines but with another monitor. Until now it is the only parameter which may predict return of spontaneous circulation. Because of this, researchers want to measure both with the same device, which gives the investigators the opportunity and advantage to compare end-tidal CO2 and cerebral saturation very precisely. In this manner researchers want to investigate the predictive value of cerebral saturation and compare it end-tidal CO2.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive OHCA patients

Exclusion Criteria:

* DNR code
* no possibility to attach cerebral oxygenation sensor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pre-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Clinical parameter: return of spontaneous circulation (ROSC) by pulse check | when ROSC occurs, within 1 day
  Difference between regional cerebral saturation and end-tidal carbon dioxide in detecting return of spontaneous circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium